CLINICAL TRIAL: NCT02865005
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study Comparing Dapsone 5% Gel (SEEGPharm SA) to Aczone® and Both Active Treatments Compared to Placebo (Vehicle) in the Treatment of Acne Vulgaris
Brief Title: Trial of Dapsone 5.0% Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seegpharm S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEEG-2015-6-23
Record Dates: First submitted 2016-07-01; First posted 2016-08-12 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dapsone 5.0% Gel (Allergan) (Active Comparator): Dapsone 5.0% Gel applied twice daily for 84 days
  Interventions: Drug: Dapsone 5.0% Gel (Allergan)
- Dapsone 5.0% Gel (SEEGPharm) (Experimental): Dapsone 5.0% Gel applied twice daily for 84 days
  Interventions: Drug: Dapsone 5.0% Gel (SEEGPharm)
- Placebo (Placebo Comparator): Vehicle of Experimental Gel applied twice daily for 84 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapsone 5.0% Gel (SEEGPharm) — Topical Gel
  Other Names: Experimental Arm
  Arms: Dapsone 5.0% Gel (SEEGPharm)
Other: Placebo — Topical Gel
  Other Names: Placebo Comparator
  Arms: Placebo
Drug: Dapsone 5.0% Gel (Allergan) — Topical Gel
  Other Names: Active Comparator
  Arms: Dapsone 5.0% Gel (Allergan)

SUMMARY:
Multi-center, double-blind, randomized, placebo-controlled trial of Dapsone 5.0% Gel in the treatment of acne vulgaris.

DETAILED DESCRIPTION:
Multi-center, double-blind, randomized, placebo-controlled trial of Dapsone 5.0% Gel in the treatment of acne vulgaris for 84 days in male and female subjects age 12-40.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant females aged ≥ 12 and ≤ 40 years of age with a clinical diagnosis of acne vulgaris.
* Informed Consent/Assent: For subjects 12 to 17 years of age inclusive must have provided Institutional Review Board (IRB) approved written assent that must be accompanied by an IRB approved written consent from the subject's legally acceptable representatives (i.e., parent or guardian). In addition, all subjects or their legally acceptable representatives must sign a Health Insurance Portability and Accountability Act (HIPAA) authorization.
* On the face, subjects must have ≥ 20 inflammatory lesions (i.e., papules and pustules), AND ≥ 25 non-inflammatory lesions (open and closed comedones) AND ≤ 2 nodulocystic lesions (i.e., nodules and cysts). For the purposes of study treatment and evaluation, all lesions on the face should be counted, including those on the nose. Subjects may have acne lesions on other areas of the body (e.g., back, chest, and arms) which should be excluded from the count, treatment and the IGA evaluation.
* Subjects must have an acne severity grade of 3 or 4 per the IGA
* Subjects must be willing to refrain from using all other topical acne medications or antibiotics during the 12-week treatment period other than the study drug.

Exclusion Criteria:

* Prior or current concomitant therapies that would interfere with assessments in the study.
* Prior or current concomitant therapies skin conditions that would interfere with assessments in the study.
* Prior, current or planned procedures that would interfere with assessments in the study.
* Current or planned activities that would interfere with assessment in the study.
* Subjects who have a Baseline local skin site reaction score of 3 [severe (marked/intense)] for any signs and/or symptoms of irritation as scored using the local skin site reaction scores.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2361 (Actual)
Dates: Start 2016-02; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Comparisons of Active Products: Mean percent change in the inflammatory lesion (papules and pustules) counts and non-inflammatory lesion (open and closed comedones) counts | Treatment Days: 84 days of dosing
  To compare Dapsone 5% Gel (SEEGPharm) to Aczone® (Allergan's Dapsone 5% Gel) to the Placebo-Vehicle control with respect to the mean percent change in the inflammatory lesion (papules and pustules) counts and non-inflammatory lesion (open and closed comedones) counts, from Baseline (Visit 1/ Day1) to End-of-Treatment (EOT)

SECONDARY OUTCOMES:
Clinical Success: Proportion of subjects with a clinical response of "success" | 12 Weeks
  To evaluate as the proportion of subjects with a clinical response of "success" at Week 12.

OTHER OUTCOMES:
Safety Outcomes: Incidence of Adverse Events | Baseline (Day 1) to Week 12 (Day 85)
  Analysis of the incidence of Adverse Events from Baseline (Day 1) to Week 12 (Day 85)
Safety Outcomes: Change in Vital Signs | Baseline (Day 1) to Week 12 (Day 85)
  Clinically Significant Changes in Body temperature (oral), pulse rate (sitting), blood pressure (sitting systolic and diastolic) from Baseline (Day 1) to Week 12 (Day 85)
Safety Outcomes: Local Skin/Application Site Reaction Scores | Baseline (Day 1) to Week 12 (Day 85)
  Application (local skin) sites will be assessed at each visit and scored using the local skin site reaction scores (0=Absent, 1=Mild, 2=Moderate, 3=Severe) for the following signs and symptoms of irritation: erythema, dryness, burning/stinging, erosion, edema, pain, and itching, for comparisons between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Lewis, MS, Study Director — Catawba Clinical Research
Locations (33):
- United States (32):
  - Catawba Clinical Research, Encino, California
  - Catawba Clinical Research, Fullerton, California
  - Catawba Clinical Research, La Mesa, California
  - Catawba Clinical Research, Los Angeles, California
  - Catawba Clinical Research, Sherman Oaks, California
  - Catawba Clinical Research, Temecula, California
  - Catawba Clinical Research, Boca Raton, Florida
  - Catawba Clinical Research, Brandon, Florida
  - Catawba Clinical Research, Hialeah, Florida
  - Catawba Clinical Research, Miami, Florida
  - Catawba Clinical Research, Miramar, Florida
  - Catawba Clinical Research, South Tampa, Florida
  - Catawba Clinical Research, Tampa, Florida
  - Catawba Clinical Research, Savannah, Georgia
  - Catawba Clinical Research, New Orleans, Louisiana
  - Catawba Clinical Research, Norfolk, Nebraska
  - Catawba Clinical Research, Omaha, Nebraska
  - Catawba Clinical Research, Las Vegas, Nevada
  - Catawba Clinical Research, Endwell, New York
  - Catawba Clinical Research, New York, New York
  - Catawba Clinical Research, High Point, North Carolina
  - Catawba Clinical Research, Wilmington, North Carolina
  - Catawba Clinical Research, Cincinnati, Ohio
  - Catawba Clinical Research, Jenkintown, Pennsylvania
  - Catawba Clinical Research, Upper Saint Clair, Pennsylvania
  - Catawba Clinical Research, Warminster, Pennsylvania
  - Catawba Clinical Research, Nashville, Tennessee
  - Catawba Clinical Research, Austin, Texas
  - Catawba Clinical Research, El Paso, Texas
  - Catawba Clinical Research, Mesquite, Texas
  - Catawba Clinical Research, Norfolk, Virginia
  - Catawba Clinical Research, Richland, Washington
- Catawba Clinical Research, Belize City, Belize

IPD SHARING:
Plan to Share IPD: No